CLINICAL TRIAL: NCT03096665
Title: Correlation Between the Point of Care Blood Analysis Obtained From Skin Puncture Blood and Conventional Blood Analysis Obtained From Venous and Arterial Blood
Brief Title: Effectiveness of Point of Care Blood Analysis Obtained From Skin Puncture Blood
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Changsun Kim, Assistant professor, Hanyang University
Other Study IDs: SKINFUNCTURE2017
Record Dates: First submitted 2017-03-14; First posted 2017-03-30 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Diseases; Acute Abdomen; Respiratory Disease; Renal Disease; Cerebrovascular Disorders
Keywords: venous blood; arterial blood; capillary blood
MeSH Terms: conditions — Cardiovascular Diseases; Abdomen, Acute; Respiration Disorders; Kidney Diseases; Cerebrovascular Disorders | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood test group: All patients receive the three types of blood test (venous blood test, skin puncture blood (capillary blood) test and arterial blood gas analysis
  Interventions: Diagnostic Test: blood test

INTERVENTIONS:
Diagnostic Test: blood test — Point of care blood analysis obtained from skin puncture

SUMMARY:
This study aimed to evaluate the correlation between the point of care blood analysis obtained from skin puncture blood and conventional blood analysis obtained from venous and arterial blood.

ELIGIBILITY:
Inclusion Criteria:

* The patients who simultaneously require the venous blood test, skin puncture blood test and arterial blood gas analysis

Exclusion Criteria:

* Unstable patients
* Patients receiving the medications affecting the results of blood analysis.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who require the blood test (venous blood test, skin puncture blood test and arteria blood gas analysis) of the patients presenting to the emergency department during the study period
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-09-30 (Estimated); Study Completion 2017-09-30 (Estimated)

PRIMARY OUTCOMES:
Blood analysis between capillary blood, venous blood and arterial blood | within 1 hour
  Primary outcome
  1. Correlation of blood concentration between skin puncture blood and venous blood
     * variables Na+ (mmol/L) K+ (mmol/L) Ca++ (mmol/L) Hct (%) Glucose (mg/dl) Creatinine (mg/dl) Cl- (mmol/L)
  2. Correlation of blood concentration between skin puncture blood and arterial blood
     * variables pH pCO2 (mmHg) pO2 (mmHg) HCO3 (mmol/L) Lactate (mmol/L)
  Spearman correlation rank test will be performed to show the agreement of two methods in each value.
  We will show the correlation coefficient for all values. Ex) The correlation coefficient of Na+, K+, Ca2+, Hct, glucose, creatinine and Cl- are ___, ___, ___, ___, ___, ___, ___, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang university guri hospital, Department of emergency medicine, Guri-si, GyeongGido, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kupke IR, Kather B, Zeugner S. On the composition of capillary and venous blood serum. Clin Chim Acta. 1981 May 5;112(2):177-85. doi: 10.1016/0009-8981(81)90376-4. PMID 7237825
- [Result] Sobiech P, Pomianowski A, Stopyra A, Kuleta Z, Zbanyszek M, Procajlo A, Rajski K. Acid-base balance parameters and ionic composition of arterial, venous and capillary blood in goats. Pol J Vet Sci. 2004;7(2):117-21. PMID 15230543
- [Result] Blumenfeld TA, Hertelendy WG, Ford SH. Simultaneously obtained skin-puncture serum, skin-puncture plasma, and venous serum compared, and effects of warming the skin before puncture. Clin Chem. 1977 Sep;23(9):1705-10. PMID 890915
- [Result] Falch DK. Clinical chemical analyses of serum obtained from capillary versus venous blood, using Microtainers and Vacutainers. Scand J Clin Lab Invest. 1981 Feb;41(1):59-62. doi: 10.3109/00365518109092015. PMID 7256193